CLINICAL TRIAL: NCT00640887
Title: Pharmacokinetics of Rifabutin Combined With Antiretroviral Therapy in the Treatment of Tuberculosis Patient With HIV Infection in South Africa: A Phase II Trial
Brief Title: Pharmacokinetics of Rifabutin Combined With Antiretroviral Therapy in Patients With TB/HIV Co-infection in South Africa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Claire Rekacewicz, French National Agency for Research on AIDS and Viral Hepatitis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANRS12150a
Record Dates: First submitted 2008-02-06; First posted 2008-03-21 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: HIV Infections; Tuberculosis
Keywords: HIV; Tuberculosis; Rifabutin; Pharmacokinetics; South Africa
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Rifabutin; efavirenz; Nevirapine; Lopinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): RBT associated with EFV based ART
  Interventions: Drug: rifabutin in combination with efavirenz
- 2 (Experimental): RBT associated with NVP based ART
  Interventions: Drug: rifabutin in combination with nevirapine
- 3 (Experimental): RBT associated with LPV/r based ART
  Interventions: Drug: rifabutin in combination with lopinavir/ritonavir

INTERVENTIONS:
Drug: rifabutin in combination with efavirenz — Ia. arm 1a:
  D4T/3TC/EFV(600mg)+INH/Rifabutin(450 mg OD 4 wks switch to 600 mg OD 4 wks);
  Ib. arm 1b:
  D4T/3TC/EFV(600mg)+INH/Rifabutin(600 mg OD 4 wks switch to 450 mg OD 4 wks);
  Arms: 1
Drug: rifabutin in combination with nevirapine — IIa. arm 2a:
  D4T/3TC/NVP(200mg)+INH/Rifabutin(300 mg OD 4 wks switch to 450 mg OD 4 wks);
  IIb. arm 2b :
  D4T/3TC/NVP(200mg)+INH/Rifabutin(450 mg OD 4 wks switch to 300 mg OD 4 wks);
  Arms: 2
Drug: rifabutin in combination with lopinavir/ritonavir — IIIa. arm 3a :
  D4T/3TC/LPV/r(2 tabs BD)+INH/Rifabutin(150 mg TPW 4 wks switch to 150 mg OD 4 wks);
  IIIb. arm 3b:
  D4T/3TC/LPV/r(2 tabs BD)+INH/Rifabutin(150 mg OD 4 wks switch to 150 mg TPW 4 wks).
  Arms: 3

SUMMARY:
The overall aim of the project is to evaluate rifabutin (RBT) as a replacement for rifampicin (RMP), for the combined treatment of tuberculosis and HIV infection. RBT represents an alternative to RMP for HIV infected patients as its half-life is longer and the enzymatic induction effect appears to be less important on the associated antiretroviral therapy (ART) drugs.

This phase II trial is to determine precisely the pharmacokinetics parameters of RBT in combination with different ART regimens in Vietnamese HIV infected patients with pulmonary tuberculosis, in order to define optimal doses that will be further tested in a larger phase III trial comparing safety, tolerability and efficacy of RBT and RMP regimens.

DETAILED DESCRIPTION:
Patients will be offered to participated in the study after the first 6 weeks of the nationally recommended TB treatment. All the enrolled patients will be switched to rifabutin and randomized, two weeks later, to one of the three study ARV regimens. The RBT doses will be then adapted to the allocated ARV regimen according to a cross over scheme. Three full pharmacokinetics profile will be performed at different time point : before initiation of ARV, after one month of the first RFB dosage and one month after the second RFB dosage.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary tuberculosis (proven by AFB positive sputum or culture)
* Having completed and adhered to 6 wks of intensive phase TB chemotherapy
* Positive HIV antibody and CD4 count >50 /mm3 and <=200
* Weight > 50 kg
* No ART in the preceding 3 months
* No more than 2 weeks or ART previously
* No grade 3 or 4 clinical or laboratory findings
* Negative pregnancy test and appropriate contraceptive measures during the duration of the trial for female of childbearing age
* Having a firm home address that is readily accessible
* Karnofsky score>=80%

Exclusion Criteria:

* History of TB within the 3 years preceding the presenting episode of TB
* Previous treatment for MDR TB
* Concomitant OI requiring additional anti-infectious treatment
* Formal contraindication to any drug used in the trial
* Diabetes mellitus requiring drug treatment
* Recreational drug or alcohol abuse
* History of drug hypersensitivity to TB or related medications
* Interrupted TB therapy for more than 1 week
* Less than 90% adherent to first 6 weeks of intensive phase chemotherapy
* Mental illness that could impair ability to give informed consent or result in poor adherence to trial protocol and therapy
* Neutropenia <1200 /L, anaemia <6.8 g/dL, liver function test > grade 2
* Requiring concomitant medications that may potentially interact with study drugs
* Pregnant or lactating women
* Karnofsky score >80%
* Any condition rendering the patient unable to understand the nature, scope, and possible consequences of thes study and to provide consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of rifabutine measured (a)before introduction of ART;(b)after ART initiation (two different doses of RBT in combination with efavirenz, nevirapine or lopinavir/ritonavir) | 2, 6 and 10 weeks after randomisation

SECONDARY OUTCOMES:
Area under the curve (AUC) of efavirenz, nevirapine and lopinavir/ritonavir in combination with two doses of rifabutine | 6 and 10 weeks after randomisation
Safety : proportion of patients with grade 3 and grade 4 adverse events | through out the trial

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D Harries, MD, PhD, Principal Investigator — The international Union Against Tuberculosis and Lung Diseases (IUATLD), Paris, France; Alexander PYM, MD, Principal Investigator — Medical Research Council, South Africa
Locations (1):
- Unit for Clinical and Biomedical TB Research (Medical Research Council), Durban, South Africa

REFERENCES:
- [Derived] Hennig S, Naiker S, Reddy T, Egan D, Kellerman T, Wiesner L, Owen A, McIlleron H, Pym A. Effect of SLCO1B1 Polymorphisms on Rifabutin Pharmacokinetics in African HIV-Infected Patients with Tuberculosis. Antimicrob Agents Chemother. 2015 Oct 19;60(1):617-20. doi: 10.1128/AAC.01195-15. Print 2016 Jan. PMID 26482301
- [Derived] Naiker S, Connolly C, Wiesner L, Kellerman T, Reddy T, Harries A, McIlleron H, Lienhardt C, Pym A. Randomized pharmacokinetic evaluation of different rifabutin doses in African HIV- infected tuberculosis patients on lopinavir/ritonavir-based antiretroviral therapy. BMC Pharmacol Toxicol. 2014 Nov 19;15:61. doi: 10.1186/2050-6511-15-61. PMID 25406657